CLINICAL TRIAL: NCT05102708
Title: Study of COVID-19 Prognostic Factors in Hospitalized Patients
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-COV-2021-75
Record Dates: First submitted 2021-10-27; First posted 2021-11-01 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: COVID-19
Keywords: Prognostic Factors; COVID-19; Hospitalization; Critical care; All-cause mortality
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Other: Prognostic factors of severe COVID-19 — prognostic factors: patients´ epidemiological characteristics (such as age, sex), comorbidities, length of hospitalization, critical care admission, treatments received, laboratory results, vital signs.

SUMMARY:
Severe COVID-19 prognostic factors have been studied worldwide throughout the pandemic, but there is considerable variability. Therefore, the investigators will summarize the identified prognostic factors in the international literature and will conduct a retrospective cohort study to identify the prognostic factors of severe COVID-19 in hospitalized patients of the Hospital de la Santa Creu i Sant Pau in Barcelona (Spain) between March 2020 and February 2021, compare them with those mentioned in the international literature and establish those most adequate to our population.

DETAILED DESCRIPTION:
Background: Spain is one of the European countries most affected by the SARS-CoV-2 pandemic, with a fatality rate of 2.2%. Faced with the significant number of patients requiring intensive care, the number of beds increased considerably in the span of 11 months to respond to the situation. There is still no drug treatment or specific prognostic factors for COVID-19 that allow its proper management.

Objective: To study the prognostic factors of severity due to COVID-19 in hospitalized patients at Hospital de la Santa Creu i Sant Pau, and their comparison with the prognostic factors identified in the literature review.

Methods: In a first phase, the published studies will be reviewed to identify the existing prognostic factors through various platforms (MEDLINE, EMBASE, Cochrane). A retrospective cohort study will subsequently be carried out to determine the patients' characteristics and to identify the prognostic factors of severity. Patients over 18 years of age, diagnosed with COVID-19 and hospitalized between March 01, 2020 and February 28, 2021 will be included. A descriptive analysis of the cohort will firstly be performed, followed by an analysis of the possible prognostic factors through bivariate tests and multivariate analyzes. The occurrence of admission to intensive care, mortality, and hospital stay > 30 days will be calculated with logistic regression (p <0.05, a = 0.05, 95% confidence interval). Finally, the prognostic factors identified in the literature review will be compared with those determined in the cohort.

ELIGIBILITY:
Inclusion Criteria:

* Equal or older than 18 years old
* Hospitalized between March 1st, 2020, and February 28th, 2021.
* Be diagnosed with COVID-19 disease

Exclusion Criteria:

* Underaged patients
* > 16h stay in the Emergency Unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult COVID-19 patients hospitalized at the San Pau Hospital of Barcelona between March 2020 and February 2021.
Sampling Method: Non-Probability Sample
Enrollment: 3725 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-28 (Actual)

PRIMARY OUTCOMES:
All cause mortality | one year
  All cause mortality of COVID-19 inpatients
Critical care admission | one year
  Critical care admission of COVID-19 inpatients
Length of stay | one year
  length of hospital stay equal or longer than 30 days
30-day all cause mortality | one year
  30-day all cause mortality of COVID-19 inpatients

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Puig, MD, PhD, MSC, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cevik M, Tate M, Lloyd O, Maraolo AE, Schafers J, Ho A. SARS-CoV-2, SARS-CoV, and MERS-CoV viral load dynamics, duration of viral shedding, and infectiousness: a systematic review and meta-analysis. Lancet Microbe. 2021 Jan;2(1):e13-e22. doi: 10.1016/S2666-5247(20)30172-5. Epub 2020 Nov 19. PMID 33521734
- [Background] Wang Y, Tian H, Zhang L, Zhang M, Guo D, Wu W, Zhang X, Kan GL, Jia L, Huo D, Liu B, Wang X, Sun Y, Wang Q, Yang P, MacIntyre CR. Reduction of secondary transmission of SARS-CoV-2 in households by face mask use, disinfection and social distancing: a cohort study in Beijing, China. BMJ Glob Health. 2020 May;5(5):e002794. doi: 10.1136/bmjgh-2020-002794. PMID 32467353
- [Background] Kronbichler A, Kresse D, Yoon S, Lee KH, Effenberger M, Shin JI. Asymptomatic patients as a source of COVID-19 infections: A systematic review and meta-analysis. Int J Infect Dis. 2020 Sep;98:180-186. doi: 10.1016/j.ijid.2020.06.052. Epub 2020 Jun 17. PMID 32562846
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Nussbaumer-Streit B, Mayr V, Dobrescu AI, Chapman A, Persad E, Klerings I, Wagner G, Siebert U, Christof C, Zachariah C, Gartlehner G. Quarantine alone or in combination with other public health measures to control COVID-19: a rapid review. Cochrane Database Syst Rev. 2020 Apr 8;4(4):CD013574. doi: 10.1002/14651858.CD013574. PMID 32267544
- [Background] Chu DK, Akl EA, Duda S, Solo K, Yaacoub S, Schunemann HJ; COVID-19 Systematic Urgent Review Group Effort (SURGE) study authors. Physical distancing, face masks, and eye protection to prevent person-to-person transmission of SARS-CoV-2 and COVID-19: a systematic review and meta-analysis. Lancet. 2020 Jun 27;395(10242):1973-1987. doi: 10.1016/S0140-6736(20)31142-9. Epub 2020 Jun 1. PMID 32497510
- [Background] Piechotta V, Chai KL, Valk SJ, Doree C, Monsef I, Wood EM, Lamikanra A, Kimber C, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2020 Jul 10;7(7):CD013600. doi: 10.1002/14651858.CD013600.pub2. PMID 32648959
- [Background] Jain V, Yuan JM. Predictive symptoms and comorbidities for severe COVID-19 and intensive care unit admission: a systematic review and meta-analysis. Int J Public Health. 2020 Jun;65(5):533-546. doi: 10.1007/s00038-020-01390-7. Epub 2020 May 25. PMID 32451563
- [Background] Zhou Y, Yang Q, Chi J, Dong B, Lv W, Shen L, Wang Y. Comorbidities and the risk of severe or fatal outcomes associated with coronavirus disease 2019: A systematic review and meta-analysis. Int J Infect Dis. 2020 Oct;99:47-56. doi: 10.1016/j.ijid.2020.07.029. Epub 2020 Jul 25. PMID 32721533
- [Background] Hatmi ZN. A Systematic Review of Systematic Reviews on the COVID-19 Pandemic. SN Compr Clin Med. 2021;3(2):419-436. doi: 10.1007/s42399-021-00749-y. Epub 2021 Jan 26. PMID 33521564
- [Background] Reddy RK, Charles WN, Sklavounos A, Dutt A, Seed PT, Khajuria A. The effect of smoking on COVID-19 severity: A systematic review and meta-analysis. J Med Virol. 2021 Feb;93(2):1045-1056. doi: 10.1002/jmv.26389. Epub 2020 Aug 13. PMID 32749705
- [Background] Moreno G, Carbonell R, Bodi M, Rodriguez A. Systematic review of the prognostic utility of D-dimer, disseminated intravascular coagulation, and anticoagulant therapy in COVID-19 critically ill patients. Med Intensiva (Engl Ed). 2021 Jan-Feb;45(1):42-55. doi: 10.1016/j.medin.2020.06.006. Epub 2020 Jun 17. PMID 32646669
- [Background] Lazarus G, Audrey J, Wangsaputra VK, Tamara A, Tahapary DL. High admission blood glucose independently predicts poor prognosis in COVID-19 patients: A systematic review and dose-response meta-analysis. Diabetes Res Clin Pract. 2021 Jan;171:108561. doi: 10.1016/j.diabres.2020.108561. Epub 2020 Dec 9. PMID 33310127
- [Background] Martha JW, Wibowo A, Pranata R. Prognostic value of elevated lactate dehydrogenase in patients with COVID-19: a systematic review and meta-analysis. Postgrad Med J. 2022 Jun;98(1160):422-427. doi: 10.1136/postgradmedj-2020-139542. Epub 2021 Jan 15. PMID 33452143
- [Background] Martha JW, Wibowo A, Pranata R. Hypocalcemia is associated with severe COVID-19: A systematic review and meta-analysis. Diabetes Metab Syndr. 2021 Jan-Feb;15(1):337-342. doi: 10.1016/j.dsx.2021.01.003. Epub 2021 Jan 18. PMID 33493853
- [Background] Chocron R, Galand V, Cellier J, Gendron N, Pommier T, Bory O, Khider L, Trimaille A, Goudot G, Weizman O, Alsac JM, Geneste L, Schmeltz A, Panagides V, Philippe A, Marsou W, Ben Abdallah I, Deney A, El Batti S, Attou S, Juvin P, Delmotte T, Messas E, Pezel T, Planquette B, Duceau B, Gaussem P, Sutter W, Sanchez O, Waldman V, Diehl JL, Mirault T, Bonnet G, Cohen A, Smadja DM; Critical COVID-19 France Investigators. Anticoagulation Before Hospitalization Is a Potential Protective Factor for COVID-19: Insight From a French Multicenter Cohort Study. J Am Heart Assoc. 2021 Apr 20;10(8):e018624. doi: 10.1161/JAHA.120.018624. Epub 2021 Feb 8. PMID 33550816
- [Background] Nugroho J, Wardhana A, Maghfirah I, Mulia EPB, Rachmi DA, A'yun MQ, Septianda I. Relationship of D-dimer with severity and mortality in SARS-CoV-2 patients : A meta-analysis. Int J Lab Hematol. 2021 Feb;43(1):110-115. doi: 10.1111/ijlh.13336. Epub 2020 Sep 15. PMID 32931146
- [Background] Thachil J, Tang N, Gando S, Falanga A, Cattaneo M, Levi M, Clark C, Iba T. ISTH interim guidance on recognition and management of coagulopathy in COVID-19. J Thromb Haemost. 2020 May;18(5):1023-1026. doi: 10.1111/jth.14810. Epub 2020 Apr 27. No abstract available. PMID 32338827
- [Background] Elavarasi A, Prasad M, Seth T, Sahoo RK, Madan K, Nischal N, Soneja M, Sharma A, Maulik SK, Shalimar, Garg P. Chloroquine and Hydroxychloroquine for the Treatment of COVID-19: a Systematic Review and Meta-analysis. J Gen Intern Med. 2020 Nov;35(11):3308-3314. doi: 10.1007/s11606-020-06146-w. Epub 2020 Sep 3. PMID 32885373
- [Background] Cavalcanti AB, Zampieri FG, Rosa RG, Azevedo LCP, Veiga VC, Avezum A, Damiani LP, Marcadenti A, Kawano-Dourado L, Lisboa T, Junqueira DLM, de Barros E Silva PGM, Tramujas L, Abreu-Silva EO, Laranjeira LN, Soares AT, Echenique LS, Pereira AJ, Freitas FGR, Gebara OCE, Dantas VCS, Furtado RHM, Milan EP, Golin NA, Cardoso FF, Maia IS, Hoffmann Filho CR, Kormann APM, Amazonas RB, Bocchi de Oliveira MF, Serpa-Neto A, Falavigna M, Lopes RD, Machado FR, Berwanger O; Coalition Covid-19 Brazil I Investigators. Hydroxychloroquine with or without Azithromycin in Mild-to-Moderate Covid-19. N Engl J Med. 2020 Nov 19;383(21):2041-2052. doi: 10.1056/NEJMoa2019014. Epub 2020 Jul 23. PMID 32706953
- See also: World Health Organization — https://www.who.int/publications/journals/bulletin
- See also: COVID-19: timeline of WHO action — https://www.who.int/es/news/item/27-04-2020-who-timeline---covid-19
- See also: World Health Organization - COVID-19 Weekly Epidemiological Update — https://www.who.int/docs/default-source/coronaviruse/situation-reports/weekly_epidemiological_update_22.pdf
- See also: WHO Coronavirus (COVID-19) Dashboard — https://covid19.who.int/
- See also: COVID-19 - UpToDate — https://www.uptodate.com/contents/covid-19-epidemiology-virology-and-prevention
- See also: Actualización de la situación epidemiológica de las variantes de SARS-CoV-2 de preocupación (VOC) e interés (VOI) en salud pública en España — https://www.mscbs.gob.es/profesionales/saludPublica/ccayes/alertasActual/nCov/documentos/COVID19_Actualizacion_variantes_20210906.pdf
- See also: John Hopkins Coronavirus Resource Center — https://coronavirus.jhu.edu/map.html
- See also: European Centre for Disease Prevention and Control (ECDC) COVID-19 situation update worldwide — https://www.ecdc.europa.eu/en/geographical-distribution-2019-ncov-cases
- See also: European Centre for Disease Prevention and Control (ECDC) COVID-19 situation update for the EU/EEA — https://www.ecdc.europa.eu/en/cases-2019-ncov-eueea
- See also: John Hopkins Coronavirus Resource Center - Mortality Analyses — https://coronavirus.jhu.edu/data/mortality
- See also: Generalitat de Catalunya COVID-19 Data — https://dadescovid.cat/
- See also: Public Health Agency of Barcelona - COVID-19 Data — https://www.aspb.cat/documents/vigilanciacovid19-dades/
- See also: Digital Economy article — https://www.economiadigital.es/politica/cataluna-tiene-el-58-de-las-camas-uci-con-enfermos-de-covid-19.html
- See also: WHO Corticosteroids for COVID-19 — https://www.who.int/publications/i/item/WHO-2019-nCoV-Corticosteroids-2020.1